CLINICAL TRIAL: NCT01448473
Title: Is a Two-Film Skull X-ray Series as Sensitive as a Four-Film Series in the Diagnosis of Skull Fractures in Paediatric Patients With Minor Head Trauma?
Brief Title: Is a Two-Film Skull X-ray Series as Sensitive as a Four-Film Series in the Diagnosis of Skull Fractures in Paediatric Patients
Acronym: 4vs2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Jocelyn Gravel, MD, St. Justine's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 4vs2
Record Dates: First submitted 2011-10-05; First posted 2011-10-07 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Head Trauma
Keywords: Head trauma; Children; Radiography
MeSH Terms: conditions — Craniocerebral Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 4 views radiograph serie (Experimental): The 4-film series will include the following views: anterior-posterior; one lateral; Waters, and Townes views.
  Interventions: Other: 4-views series
- 2-view radiography serie (Active Comparator): The 2-film series will include the following views: anterior-posterior and one lateral.
  Interventions: Other: 2-views serie

INTERVENTIONS:
Other: 4-views series — The 4-film series will include the following views: anterior-posterior; one lateral; Waters, and Townes views.
  Arms: 4 views radiograph serie
Other: 2-views serie — The 2-film series will include the following views: anterior-posterior and one lateral.
  Arms: 2-view radiography serie

SUMMARY:
Minor head injuries are a common presenting complaint in the pediatric emergency department. Skull x-rays are a useful tool in the evaluation of paediatric patients with a history of minor head trauma. However, there exists ongoing controversy regarding the ideal number of views that should be obtained in a skull series. This study aims to determine if there is a significant difference in the diagnostic accuracy of skull x-rays in the diagnosis of fracture in paediatric minor head trauma patients when a 2-film series as opposed to a 4-film series is provided to participating pediatric emergency physicians.

DETAILED DESCRIPTION:
Minor head injuries are a common presenting complaint in the pediatric emergency department. Skull x-rays are a useful tool in the evaluation of paediatric patients with a history of minor head trauma. However, there exists ongoing controversy regarding the ideal number of views that should be obtained in a skull series. This study aims to determine if there is a significant difference in the diagnostic accuracy of skull x-rays in the diagnosis of fracture in paediatric minor head trauma patients when a 2-film series as opposed to a 4-film series is provided to participating pediatric emergency physicians.

This will be a prospective, crossover experimental study evaluating the equivalency in sensitivity and specificity of a 2-film series versus a 4-film series in the diagnosis of skull fracture associated with minor head injuries in children.

The study will involve 10 pediatric emergency physicians who will evaluate two modules of 100 series of radiography.

In order to do so, he or she will be given two work modules. Each module will contain the randomized and anonymous x-rays of the same 50 cases and 50 controls mounted on power point slides. Among the 50 cases, the evaluation sequence will be randomized such that 25 cases will be evaluated with the 2-film series in the first module and the 4-film series in the second module while the other 25 cases will evaluated in the reverse order. The same procedure will be used for randomizing the evaluation sequence of the 50 controls.

The primary outcomes will be the overall sensitivity and specificity of pediatric emergency medicine physicians for the detection of skull fractures using two evaluation methods: one in which they are presented with a skull series that has 2 views and another in which they are presented with a standard 4-view series.

ELIGIBILITY:
Inclusion Criteria:

* Children who had a radiography for head trauma

Exclusion Criteria:

* None

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Sensitivity
  The sensitivity is a simple proportion and will be measured by dividing the number of cases that were classified as positive for fracture by the total number of cases.
Specificity
  The specificity will be measured by dividing the number of x-rays of controls in which x-rays were read as negative by the total number of x-rays of controls.

SECONDARY OUTCOMES:
Individual sensitivity
  The sensitivity of individual participants in the detection of skull fracture will be calculated.
Individual specificity
  The specificity of individual participants in the detection of skull fracture will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyn Gravel, MD, Principal Investigator — Sainte-Justine Hospital
Locations (1):
- Sainte-Justine Hospital, Montreal, Quebec, Canada